CLINICAL TRIAL: NCT03407729
Title: Structure & Function of Dopaminergic Brain Networks Following Postnatally-Occurring Hypoxic Insults
Brief Title: Measuring Brain Activity of School Age Children
Status: Completed | Type: Observational
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Michael J. Decker, Associate Professor, Case Western Reserve University
Other Study IDs: 12266077; 05-17-23 (Other: UHCMC IRB)
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Results first posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Perinatal Hypoxia; Dopamine; Neurobehavioral Manifestations
Keywords: Hypoxia, Brain; Neural networks; Magnetic Resonance Imaging
MeSH Terms: conditions — Neurobehavioral Manifestations; Hypoxia, Brain | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — MRI neuroimages
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post-hypoxic former preterm: Born in the years 2005-2009 with birth gestational age between 23-28 weeks and birth weight appropriate for gestational age (AGA). Part of a research cohort with available oxygen saturation level data recorded continuously from the first day of life to 8 weeks postnatal age (n=11).Children will undergo Magnetic Resonance Imaging and Cognitive Performance Testing.
  Interventions: Other: Magnetic Resonance Imaging; Other: Cognitive Performance Testing
- Healthy term-born children: Born in the years 2005-2009 with birth gestational age ≥ 38 weeks gestation and birth weight appropriate for term gestation (n=10) matched by age/sex/race to participating cohort children with no history of respiratory difficulty suggesting hypoxic exposure. Children will undergo Magnetic Resonance Imaging and Cognitive Performance Testing.
  Interventions: Other: Magnetic Resonance Imaging; Other: Cognitive Performance Testing

INTERVENTIONS:
Other: Magnetic Resonance Imaging — MRI uses a strong magnetic field and radio waves to create detailed images of the brain while the person's head is positioned inside a round tunnel.
  Other Names: T-1 MPRAGE; fMRI-BOLD
Other: Cognitive Performance Testing — For the Grooved Pegboard task: After the MRI scan, children will be timed as they place pegs into holes with randomly positioned slots.
  Other Names: Grooved pegboard task

SUMMARY:
This observational study will investigate whether differences in birth events and oxygen levels during the newborn period affects the brain activity of children during the middle childhood years.

DETAILED DESCRIPTION:
The investigators will conduct an observational study comparing two groups of children to determine whether differences in birth events and oxygen levels during the newborn period lead to structural and functional impairment within the brain's dopaminergic pathways and the cortical regions innervated by those pathways. The dopaminergic system is involved in modulating motor control and cognitive function.

Using magnetic resonance diffusion tensor imaging, structural integrity of dopaminergic circuits will be quantified and compared in post-hypoxic former preterm children versus healthy control children born at term closely matched by age/sex/race.

Functional activity during executive function tasks will be quantified and compared in post-hypoxic former preterm children versus healthy control children born at term using functional magnetic resonance imaging-blood oxygen level dependent (fMRI-BOLD). Assessment of motor function (grooved pegboard task) will also be performed.

ELIGIBILITY:
Inclusion Criteria:

1. For Study Group Children: Birth gestational age between 23-28 weeks and birth weight appropriate for gestational age (AGA) with available oxygen saturation level data recorded continuously from the first day of life to 8 weeks postnatal age (n=11)
2. For Healthy Control Children: Birth gestational age ≥ 38 weeks gestation and birth weight appropriate for term gestation (n=10) matched by age/sex/race to participating cohort children.
3. Born in years 2005-2009 (age range will be 8-15 years during the funding period)
4. Ability of the child to provide assent, with the parent/legal guardian able to provide written informed consent for study procedures.
5. Sensory and motor capability to complete study tasks (i.e. Grooved Pegboard test). Mental Development index must be > 80 at 2-year-old follow-up for preterm cohort.

Exclusion Criteria:

1. Past history of concussion requiring medical treatment to avoid confounding of MRI data
2. Current diagnosis of autism.
3. Child who suffers from claustrophobia (per parent report).
4. Unable to participate in neuroimaging due to claustrophobia, or medical contraindication to MRI including any implanted medical device, dental braces, surgical clips for aneurysms in the head, heart valve prostheses, electrodes or other metallic objects, pregnancy.
5. Healthy control children who were treated in the Neonatal ICU in the newborn period for breathing difficulties.
6. Healthy control children who were hospitalized for breathing problems in the first 3 months of infancy.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Study Group Children (n=11) will be drawn from a cohort currently maintained by the investigators.
  Healthy Control Children will be recruited using various strategies: (1) study flyers given to the parents of the prematurely born cohort children to pass along to parents of other children with ages similar to their own child. (2) study flyers posted in the hospital's primary care pediatric clinics asking interested children/families to contact us to learn more about the study; (3) study flyers distributed by professional colleagues/pediatric physicians to potential candidate children/families meeting study inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Decker, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
Because this is a vulnerable population and a small sample size from a known cohort of children, it is unclear of the institutional requirements for sharing individual participant data in any format other than peer-reviewed publications. The investigators will make datasets from this study available upon completion of the study. Those who are interested will submit a brief research plan to the Principal Investigators. Qualified investigators whose research question can be appropriately addressed by the requested dataset will be invited to discuss their plan and finalize details with the investigators via phone or in person.

REFERENCES:
- [Background] Poets CF, Samuels MP, Southall DP. Epidemiology and pathophysiology of apnoea of prematurity. Biol Neonate. 1994;65(3-4):211-9. doi: 10.1159/000244055. PMID 8038285
- [Background] Huppi PS, Murphy B, Maier SE, Zientara GP, Inder TE, Barnes PD, Kikinis R, Jolesz FA, Volpe JJ. Microstructural brain development after perinatal cerebral white matter injury assessed by diffusion tensor magnetic resonance imaging. Pediatrics. 2001 Mar;107(3):455-60. doi: 10.1542/peds.107.3.455. PMID 11230582
- [Background] Inder TE, Volpe JJ. Mechanisms of perinatal brain injury. Semin Neonatol. 2000 Feb;5(1):3-16. doi: 10.1053/siny.1999.0112. PMID 10802746
- [Background] Poets CF, Roberts RS, Schmidt B, Whyte RK, Asztalos EV, Bader D, Bairam A, Moddemann D, Peliowski A, Rabi Y, Solimano A, Nelson H; Canadian Oxygen Trial Investigators. Association Between Intermittent Hypoxemia or Bradycardia and Late Death or Disability in Extremely Preterm Infants. JAMA. 2015 Aug 11;314(6):595-603. doi: 10.1001/jama.2015.8841. PMID 26262797
- [Background] Janvier A, Khairy M, Kokkotis A, Cormier C, Messmer D, Barrington KJ. Apnea is associated with neurodevelopmental impairment in very low birth weight infants. J Perinatol. 2004 Dec;24(12):763-8. doi: 10.1038/sj.jp.7211182. PMID 15329741
- [Background] Perna R, Cooper D. Perinatal cyanosis: long-term cognitive sequelae and behavioral consequences. Appl Neuropsychol Child. 2012;1(1):48-52. doi: 10.1080/09084282.2011.643946. PMID 23428277
- [Background] Smith TF, Schmidt-Kastner R, McGeary JE, Kaczorowski JA, Knopik VS. Pre- and Perinatal Ischemia-Hypoxia, the Ischemia-Hypoxia Response Pathway, and ADHD Risk. Behav Genet. 2016 May;46(3):467-77. doi: 10.1007/s10519-016-9784-4. Epub 2016 Feb 26. PMID 26920003
- [Background] Decker MJ, Hue GE, Caudle WM, Miller GW, Keating GL, Rye DB. Episodic neonatal hypoxia evokes executive dysfunction and regionally specific alterations in markers of dopamine signaling. Neuroscience. 2003;117(2):417-25. doi: 10.1016/s0306-4522(02)00805-9. PMID 12614682
- [Background] Decker MJ, Jones KA, Solomon IG, Keating GL, Rye DB. Reduced extracellular dopamine and increased responsiveness to novelty: neurochemical and behavioral sequelae of intermittent hypoxia. Sleep. 2005 Feb;28(2):169-76. doi: 10.1093/sleep/28.2.169. PMID 16171240
- [Background] Decker MJ, Jones KA, Keating GL, Rye DB. Postnatal hypoxia evokes persistent changes within the male rat's dopaminergic system. Sleep Breath. 2018 May;22(2):547-554. doi: 10.1007/s11325-017-1558-6. Epub 2017 Aug 22. PMID 28828549
- [Background] Rocha-Ferreira E, Hristova M. Plasticity in the Neonatal Brain following Hypoxic-Ischaemic Injury. Neural Plast. 2016;2016:4901014. doi: 10.1155/2016/4901014. Epub 2016 Mar 7. PMID 27047695
- [Background] Nyakas C, Buwalda B, Luiten PG. Hypoxia and brain development. Prog Neurobiol. 1996 May;49(1):1-51. doi: 10.1016/0301-0082(96)00007-x. PMID 8817697
- [Background] Stollstorff M, Foss-Feig J, Cook EH Jr, Stein MA, Gaillard WD, Vaidya CJ. Neural response to working memory load varies by dopamine transporter genotype in children. Neuroimage. 2010 Nov 15;53(3):970-7. doi: 10.1016/j.neuroimage.2009.12.104. Epub 2010 Jan 4. PMID 20053379
- [Background] Langer N, von Bastian CC, Wirz H, Oberauer K, Jancke L. The effects of working memory training on functional brain network efficiency. Cortex. 2013 Oct;49(9):2424-38. doi: 10.1016/j.cortex.2013.01.008. Epub 2013 Jan 31. PMID 23489778
- [Background] Allin MP, Kontis D, Walshe M, Wyatt J, Barker GJ, Kanaan RA, McGuire P, Rifkin L, Murray RM, Nosarti C. White matter and cognition in adults who were born preterm. PLoS One. 2011;6(10):e24525. doi: 10.1371/journal.pone.0024525. Epub 2011 Oct 12. PMID 22022357
- [Background] Alexander AL, Lee JE, Lazar M, Field AS. Diffusion tensor imaging of the brain. Neurotherapeutics. 2007 Jul;4(3):316-29. doi: 10.1016/j.nurt.2007.05.011. PMID 17599699
- [Background] D'Ardenne K, McClure SM, Nystrom LE, Cohen JD. BOLD responses reflecting dopaminergic signals in the human ventral tegmental area. Science. 2008 Feb 29;319(5867):1264-7. doi: 10.1126/science.1150605. PMID 18309087
- [Background] Kim SG, Ogawa S. Biophysical and physiological origins of blood oxygenation level-dependent fMRI signals. J Cereb Blood Flow Metab. 2012 Jul;32(7):1188-206. doi: 10.1038/jcbfm.2012.23. Epub 2012 Mar 7. PMID 22395207
- [Background] Goncalves SI, de Munck JC, Pouwels PJ, Schoonhoven R, Kuijer JP, Maurits NM, Hoogduin JM, Van Someren EJ, Heethaar RM, Lopes da Silva FH. Correlating the alpha rhythm to BOLD using simultaneous EEG/fMRI: inter-subject variability. Neuroimage. 2006 Mar;30(1):203-13. doi: 10.1016/j.neuroimage.2005.09.062. Epub 2005 Nov 14. PMID 16290018
- [Background] Galan RF, Ermentrout GB, Urban NN. Efficient estimation of phase-resetting curves in real neurons and its significance for neural-network modeling. Phys Rev Lett. 2005 Apr 22;94(15):158101. doi: 10.1103/PhysRevLett.94.158101. Epub 2005 Apr 19. PMID 15904191

RESULTS

PARTICIPANT FLOW:
Groups:
- Post-hypoxic Former Preterm: Born in the years 2005-2009 with birth gestational age between 23-28 weeks and birth weight appropriate for gestational age (AGA). Part of a research cohort with available oxygen saturation level data recorded continuously from the first day of life to 8 weeks postnatal age (n=11).Children will undergo Magnetic Resonance Imaging, Electroencephalography, and Cognitive Performance Testing.
  Magnetic Resonance Imaging: MRI uses a strong magnetic field and radio waves to create detailed images of the brain while the person's head is positioned inside a round tunnel.
  Electroencephalography: EEG tracks and records brain wave patterns. A head cap with small discs and thin wires (electrodes) is placed on the scalp, and then send signals to a computer.
  Cognitive Performance Testing: For the Verbal n-back: During the fMRI scan, children will respond to a letter displayed on a small screen and indicate (by pushing a button) whether the letter shown is the same as a previously displayed letter. Children will repeat this test during the EEG.
  For the Grooved Pegboard task: After the MRI scan, children will be timed as they place pegs into holes with randomly positioned slots.
- Healthy Term-born Children: Born in the years 2005-2009 with birth gestational age ≥ 38 weeks gestation and birth weight appropriate for term gestation (n=10) matched by age/sex/race to participating cohort children with no history of respiratory difficulty suggesting hypoxic exposure. Children will undergo Magnetic Resonance Imaging, Electroencephalography, and Cognitive Performance Testing.
  Magnetic Resonance Imaging: MRI uses a strong magnetic field and radio waves to create detailed images of the brain while the person's head is positioned inside a round tunnel.
  Electroencephalography: EEG tracks and records brain wave patterns. A head cap with small discs and thin wires (electrodes) is placed on the scalp, and then send signals to a computer.
  Cognitive Performance Testing: For the Verbal n-back: During the fMRI scan, children will respond to a letter displayed on a small screen and indicate (by pushing a button) whether the letter shown is the same as a previously displayed letter. Children will repeat this test during the EEG.
  For the Grooved Pegboard task: After the MRI scan, children will be timed as they place pegs into holes with randomly positioned slots.
Period: Overall Study
Arm/Group | Post-hypoxic Former Preterm | Healthy Term-born Children
Started | 11 | 10
Completed | 9 | 7
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Unable to schedule | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Post-hypoxic Former Preterm | Healthy Term-born Children | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 7 | 16
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.15 (0.93) | 12.13 (2.06) | 11.58 (1.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 7 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 1 | 4 | 5
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 7 | 16
Birth gestation [Mean (Standard Deviation); unit: weeks] — gestational at birth (maternal pregnancy weeks completed)
  weeks | 26.11 (1.90) | 39.00 (1.00) | 31.75 (6.78)

OUTCOME MEASURES:

1. Primary Outcome: Structural Integrity of Dopaminergic Circuits
Description: Assessment of dopaminergic circuits originating in the substantia nigra pars compacta (SNpc) and ventral tegmental area (VTA). Includes right and left nucleus accumbens, right and left mamillary body, right and left hippocampus. Measured using Magnetic Resonance T1-weighted magnetization prepared rapid gradient echo (MPRAGE) scans with three-dimensional volumetrics analysis
Time Frame: 30 minutes
Population: All participants who had a usable structural magnetic resonance imaging (MRI) scan
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Post-hypoxic Former Preterm | Healthy Term-born Children
Number analyzed (Participants) | 9 | 7
mm^3
  left nucleus accumbens | 148.90 (50.12) | 175.93 (25.41)
  right nucleus accumbens | 177.25 (31.46) | 192.78 (16.48)
  left mamillary body | 89.34 (18.18) | 54.78 (18.02)
  right mamillary body | 67.78 (17.34) | 44.70 (15.03)
  left hippocampus | 2741.09 (511.83) | 3419.48 (619.00)
  right hippocampus | 3329.34 (682.48) | 4241.03 (659.36)

2. Primary Outcome: Functional Activity During Executive Function Tasks
Description: Subjects in each group were evaluated for changes in functional connectivity between the substantia nigra pars compacta (SNpc) and ventral tegmental area (VTA), as evaluated by functional magnetic resonance imaging blood oxygen level dependent (fMRI-BOLD), using whole brain analysis. The measurement is increase/decrease of MRI signal intensity in a given region, thresholded at p <0.05, summarized into a value representing 'size of region of increase' or 'size of region of decrease' after subjects' scans were combined/mapped onto a standard MNI brain. Only clusters of over 50 voxels were included, and the size of the region is reported in voxel size. The averaged brains for prematurely born fMRI was subtracted from the full term treatment for each group, and then these averaged differences were subtracted from each other. While other areas of the brain met threshold criteria in the analysis, only brain regions innervated by primary or collateral dopaminergic pathways are reported.
Time Frame: 30 minutes
Population: All participants who met criteria for a technically acceptable functional magnetic resonance imaging scan (less than 3mm movement artifact) were included in these analyses. FSL (FMRIB Software Library)-defined cluster sizes greater than 50 voxels, with p<0.05, within cognitive areas of interest are included in the outcome table. That table provides the number of voxels in clusters that showed increased or decreased connectivity.
Measure: Number; unit: Cluster size (voxels)
Arm/Group | Post-hypoxic Former Preterm | Healthy Term-born Children
Number analyzed (Participants) | 7 | 6
Cluster size (voxels)
  Left thalamus | 310 | 358
  Left middle temporal gyrus | 95 | 75
Statistical Analysis 1: Comparison: Post-hypoxic Former Preterm vs Healthy Term-born Children; Test type: Other — Using seed-based analysis with a 1) Left Thalamus seed and 2) Left Middle Temporal Gyrus seed, cluster size was set at 50 voxels and p-value was thresholded at p<0.05. This was used to compare the differences between the two study groups in terms of number of activated voxels during during cognitive testing using the N-back; p < 0.05, t-test, 2 sided — The a priori threshold for statistical significance was p<0.05 and statistical power was set at a minimum of 0.80

3. Secondary Outcome: Cognitive Performance-Fine Motor Function
Description: Measured using the grooved pegboard task (number of seconds required to place 25 pegs using the dominant hand)
Time Frame: 20 minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Post-hypoxic Former Preterm | Healthy Term-born Children
Number analyzed (Participants) | 9 | 7
seconds | 102.11 (42.77) | 82.71 (15.59)

ADVERSE EVENTS:
Time Frame: 1 week
Groups:
- Post-hypoxic Former Preterm: Born in the years 2005-2009 with birth gestational age between 23-28 weeks and birth weight appropriate for gestational age (AGA). Part of a research cohort with available oxygen saturation level data recorded continuously from the first day of life to 8 weeks postnatal age (n=11).Children will undergo Magnetic Resonance Imaging, Electroencephalography, and Cognitive Performance Testing.
  Magnetic Resonance Imaging: MRI uses a strong magnetic field and radio waves to create detailed images of the brain while the person's head is positioned inside a round tunnel.
  Cognitive Performance Testing: For the Grooved Pegboard task: After the MRI scan, children will be timed as they place pegs into holes with randomly positioned slots.
- Healthy Term-born Children: Born in the years 2005-2009 with birth gestational age ≥ 38 weeks gestation and birth weight appropriate for term gestation (n=10) matched by age/sex/race to participating cohort children with no history of respiratory difficulty suggesting hypoxic exposure. Children will undergo Magnetic Resonance Imaging, Electroencephalography, and Cognitive Performance Testing.
  Magnetic Resonance Imaging: MRI uses a strong magnetic field and radio waves to create detailed images of the brain while the person's head is positioned inside a round tunnel.
  Cognitive Performance Testing: For the Grooved Pegboard task: After the MRI scan, children will be timed as they place pegs into holes with randomly positioned slots.
Arm/Group | Post-hypoxic Former Preterm | Healthy Term-born Children
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 0/9 | 0/7

LIMITATIONS AND CAVEATS:
Insufficient numbers of children studied due to severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) pandemic research shut-down. When research protocols were permitted to resume, parents were reluctant to bring children for a voluntary research study. Data collection also terminated early for technical reasons; the magnetic resonance imaging (MRI) scanner was replaced during the pandemic shut-down with a different model that did not produce comparable results to the earlier scans.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-13): https://cdn.clinicaltrials.gov/large-docs/29/NCT03407729/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/29/NCT03407729/ICF_001.pdf